CLINICAL TRIAL: NCT02992054
Title: Randomized Controlled Trial for Assessing the Effects Resulting From an Innovative Occupational Program Using New Technologies (KODRO) on Nursing Home Residents' Quality of Life (Pilot Study)
Brief Title: An Innovative Occupational Program Using New Technologies (KODRO) Life of Nursing
Acronym: KODRO
Status: Terminated | Type: Observational
Why Stopped: The number of patients were enough for statistic treatment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9215
Record Dates: First submitted 2016-09-06; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2014-12

CONDITIONS: Home Residents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stimulating activities with the use of tactile tablet computer: Stimulating activities through the use of a tactile tablet computer. These tablets are linked to an internet-based service platform and offer a very easy and intuitive interaction for the user, even when this person is suffering from a moderate cognitive and/or physical impairment.
  Interventions: Other: stimulating activities
- Stimulating activities with usual stimulation activity program: No Stimulating activities through the use of a tactile tablet computer

INTERVENTIONS:
Other: stimulating activities
  Groups: Stimulating activities with the use of tactile tablet computer

SUMMARY:
Randomized controlled trial for assessing the effects resulting from an innovative occupational program using new technologies (KODRO) on nursing home residents' quality of life

Context : improving quality of life (QOL) for the nursing homes residents (NHR) is a national priority (2010 report from French ANESM).

DETAILED DESCRIPTION:
KODRO stimulation program makes available stimulating activities through the use of a tactile tablet computer. These tablets are linked to an internet-based service platform The project main objective is to demonstrate by way of a randomized controlled trial the significance of the improvement of residents' QOL achieved by 2 one-hour KODRO sessions per week during 6 months (KODRO nursing homes) when compared with the usual stimulation activity program (nursing homes "controls") (difference for the QOL-AD score > 2 points).At last, the objective of the study is also observational, i.e. to determine the quality of life of NHR at baseline, in its differents aspects.Subjects & methods Analysis will be conducted to compare quantitative parameters at the beginning of the trial to verify the comparability of the two groups and of the mean average change between parameters measured at baseline, 3 months, and 6 months in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents

Exclusion Criteria:

* Not able to participate in the ocupational therapy using KODRO (Demential end of life ...)

Ages: 65 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2010-12; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Quality of life: QOL-AD score: questionnaire | 6 months

SECONDARY OUTCOMES:
Different aspects of QOL score: questionnaire | 6 Months
  Measurement of apathy
  * depression
  * anxiety
  * autonomy
  * self-esteem
  * overall well-being
  * behavioral problems
  * psychotropic medication use

CONTACTS AND LOCATIONS:
Overall Officials: Hubert BLAIN, MD, PHD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: No